CLINICAL TRIAL: NCT03300427
Title: Controlled Trial on the Short-term Effects of Sacubitril/Valsartan Therapy on Cardiac Oxygen Consumption and Efficiency of Cardiac Work in Patients With NYHA II-III Heart Failure and Reduced Systolic Function Using 11C-acetate Positron Emission Tomography and Echocardiography
Brief Title: The Effects of Sacubitril/Valsartan on Cardiac Oxygen Consumption and Efficiency of Cardiac Work in Heart Failure Patients
Acronym: TurkuPET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCZ696BFI03; 2017-002113-64 (EudraCT Number)
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: Heart failure with reduced left ventricular ejection fraction; LVEF; Cardiac dysfunction; Heart muscle dysfunction; Left ventricular (LV) dilation; Left ventricular hypertrophy; HF; AHF; CHF; CCF; acute heart failure; chronic heart failure; congestive heart failure; congestive cardiac failure
MeSH Terms: conditions — Heart Failure; Dilatation, Pathologic; Hypertrophy, Left Ventricular | interventions — sacubitril; Valsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sacubitril/valsartan (Experimental): subjects received sacubitril/valsartan 100 mg orally twice daily (BID). The dose was then up-titrated to 200 mg BID (or maintained at the starting dose level, if up-titration was not possible).
  Interventions: Drug: sacubitril/valsatran; Drug: placebo to valsartan
- valsartan (Active Comparator): subjects received 80 mg orally twice daily (BID). The dose was then up-titrated to 160 mg BID (or maintained at the starting level, if up-titration was not possible)
  Interventions: Drug: valsartan; Drug: placebo to sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsatran — sacubitril/valsatran 100 or 200 mg BID
  Arms: sacubitril/valsartan
Drug: valsartan — Valsartan 80 or 160 mg BID
  Arms: valsartan
Drug: placebo to valsartan — placebo to valsartan 80 or 160 BID
  Arms: sacubitril/valsartan
Drug: placebo to sacubitril/valsartan — placebo to sacubitril/valsartan 100 or 200 mg BID
  Arms: valsartan

SUMMARY:
This is a phase IV, prospective, randomized, double-blind, double-dummy, parallel-group study.

The study assessed the effects of 6 weeks of stable sacubitril/valsartan therapy, as compared with valsartan therapy, on the efficiency of cardiac work in patients with NYHA II-III heart failure (HF) and reduced systolic function using 11C-acetate positron emission tomography (PET) and echocardiography.

DETAILED DESCRIPTION:
Subjects were randomized into valsartan or sacubitril/valsartan arms in a 1:1 ratio. Regardless of the treatment arm a subject is in, the study drug was up-titrated to the highest tolerated dose level during the scheduled study visits. The different strengths of the two study drugs were not identical in appearance so the possible dose modification(s) during the treatment period could not be performed in a blinded manner. Subjects started on valsartan 80 mg BID or sacubitril/valsartan 100 mg BID dose and there was only one scheduled up-titration visit after the randomization. Exception for this were the subjects that were on valsartan 160 mg BID dose during the run-in phase. These subjects were randomized directly to valsartan 160 mg BID or sacubitril/valsartan 100 mg BID. Subjects that were randomized to valsartan arm had similar visit after which they continued on the same dose. For subjects that were randomized from valsartan 160 mg BID to sacubitril/valsartan 100 mg BID the dose was up-titrated to 200 mg BID if clinically possible.

The total duration for each patient was planned to be about 14 weeks but could be longer if required for scheduling purposes . The longest participation, from signing of ICF until end of study, was 26 weeks.

ELIGIBILITY:
Inclusion criteria:

* 40-80 years of age
* Chronic HF with reduced EF (left ventricle EF 25-35%) and NYHA class II-III symptoms.
* Systolic BP 110-160 mm Hg
* Optimal standard HF therapy according to European Society of Cardiology (ESC) guidelines at a stable dose for at least 4 weeks before the screening visit.

Exclusion criteria:

* Estimated glomerular filtration rate (eGFR) < 45 ml/min
* Serum potassium > 5.2 mmol/l and creatinine >1.5 x ULN

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The patients who signed the ICF entered the screening/run-in period of the study. After the screening evaluations and confirmation of eligibility, the patients were allocated randomization numbers and randomized to receive the treatment assigned to each number in a blinded manner.
Groups:
- Sacubitril/Valsartan: subjects receive sacubitril/valsartan 100 mg orally twice daily (BID). The dose is then up-titrated to 200 mg BID (or maintained at the starting dose level, if up-titration is not possible).
- Valsartan: subjects receive 80 mg orally twice daily (BID). The dose is then up-titrated to 160 mg BID (or maintained at the starting level, if up-titration is not possible)
Period: Overall Study
Arm/Group | Sacubitril/Valsartan | Valsartan
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sacubitril/Valsartan | Valsartan | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (10.1) | 64.4 (7.5) | 63.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 22 | 21 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Energetic Efficiency
Description: Positron emission tomography (PET) imaging and echocardiography were performed before randomization (after a minimum of 4 weeks on stable dose of 80 mg BID or 160 mg BID of valsartan) and repeated after 6 weeks on a stable dose of either 80 mg BID or 160 mg BID of valsartan or 100 mg BID or 200 mg BID of sacubitril/valsartan.
  Cardiac efficiency was calculated based on the following formula: Myocardial efficiency = ((SBP x SV x HR)/LV mass)/Kmono Where
  * SBP : Systolic blood pressure during PET
  * SV : Stroke volume (Echocardiography)
  * HR : Heart rate
  * Kmono: Mono-exponential clearance rate (11C-acetate PET- scan)
  * LV mass: Left ventricular mass
  Visit 3 was performed after the study treatment was on a stable dose for a minimum of 6 weeks. It could be performed before or after 8 weeks, based on when the last dose modification was performed.
  No imputation of missing data was performed.
Time Frame: Baseline, Visit 3 (approximately Week 8)
Population: Full analysis set (FAS): consisted of all randomized patients who had received at least one dose of study medication in the treatment period and had at least one post-baseline assessment of any efficacy endpoints.
Measure: Mean (Standard Deviation); unit: (((mmhg x ml x bpm) /g)/(1/min))
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 27 | 28
(((mmhg x ml x bpm) /g)/(1/min))
  Baseline (Day 1) | 48621.3 (17001.4) | 50035.7 (18068.2)
  Visit 3 | 50301.0 (20842.7) | 52942.8 (19702.5)

2. Primary Outcome: Change From Baseline in Myocardial Energetic Efficiency
Description: as for outcome 1
Time Frame: Baseline, Visit 3 (approximately Week 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (((mmhg x ml x bpm) /g)/(1/min))
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 27 | 28
(((mmhg x ml x bpm) /g)/(1/min)) | 1679.8 (9282.4) | 2907.1 (11571.5)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; The study hypothesis is that short-term therapy with sacubitril/valsartan added on standard HF therapy improves cardiac efficiency in subjects with systolic HF; Test type: Superiority; p = 0.7594, ANCOVA; difference in least square means = -900.0, 95% CI 2-sided [-6781.7 to 4981.8]

3. Primary Outcome: Viable Myocardial Energetic Efficiency (Sensitivity Analysis)
Description: In addition to the derivation of the primary endpoint, an alternative formula was used, where the viable myocardial energetic efficiency was derived as:
  Viable myocardial energetic efficiency = ((SBP x SV x HR)/LV mass) / vKmono Where vKmono is the viable myocardium clearance rate. This alternative parameter was included as a sensitivity analysis to exclude possible bias related to scar tissue in patients with ischemic myopathy.
Time Frame: Baseline, Visit 3 (approximately Week 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (((mmhg x ml x bpm) /g)/(1/min))
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 27 | 28
(((mmhg x ml x bpm) /g)/(1/min))
  Baseline | 48163.0 (16719.8) | 49575.6 (18255.8)
  Visit 3 | 49914.4 (20821.2) | 52249.9 (19585.8)

4. Primary Outcome: Change From Baseline in Viable Myocardial Energetic Efficiency (Sensitivity Analysis)
Description: as for outcome 3
Time Frame: Baseline, Visit 3 (approximately Week 8)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (((mmhg x ml x bpm) /g)/(1/min))
Arm/Group | Sacubitril/Valsartan | Valsartan
Number analyzed (Participants) | 27 | 28
(((mmhg x ml x bpm) /g)/(1/min)) | 1751.4 (9098.1) | 2674.3 (11551.2)
Statistical Analysis 1: Comparison: Sacubitril/Valsartan vs Valsartan; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8422, ANCOVA; difference in least square means = -575.5, 95% CI 2-sided [-6365.5 to 5214.5]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 86 days.
Description: The occurrence of adverse events was sought by non-directive questioning of the patient at each visit during the study. Adverse events were also detected when they were volunteered by the patient during or between visits or through physical examination findings, laboratory test findings, or other assessments.
Arm/Group | Sacubitril/Valsartan | Valsartan
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/28
Other Adverse Events (participants affected / at risk) | 4/27 | 5/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sacubitril/Valsartan (N=27) | Valsartan (N=28)
Cerebrovascular accident (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sacubitril/Valsartan (N=27) | Valsartan (N=28)
Nausea (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Blood potassium increased (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT03300427/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT03300427/SAP_001.pdf